CLINICAL TRIAL: NCT00835471
Title: A Randomized Phase II Study of Erlotinib Compared to Single Agent Chemotherapy-erlotinib Combination in Pretreated Patients With Advanced NSCLC (NVALT10 Study)
Brief Title: 2nd Line Erlotinib Treatment With (Out) Chemotherapy of Advanced Non Small Cell Lung Cancer (NSCLC)
Acronym: NVALT10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dutch Society of Physicians for Pulmonology and Tuberculosis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVALT10
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung cancer; non-small-cell; erlotinib; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Erlotinib plus docetaxel (squamous cell NSCLC) or pemetrexed (non-squamous cell NSCLC)
  Interventions: Drug: erlotinib plus docetaxel or pemetrexed
- 2 (Active Comparator): Erlotinib
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib plus docetaxel or pemetrexed — non-squamous carcinoma: pemetrexed 500 mg/m2 on Day 1 plus erlotinib 150 mg/day days 2-16, every 21 days. Pemetrexed will be given for a maximum of 4 cycles. Thereafter erlotinib will be continued continuously until disease progression.
  squamous carcinoma: Docetaxel 75mg/m2 on Day 1 plus erlotinib 150mg/day days 2-16, every 21 days. Docetaxel will be given for a maximum of 4 cycles. Thereafter erlotinib will be continued continuously until disease progression.
  Other Names: Tarceva; Taxotere; Alimta
  Arms: 1
Drug: erlotinib — erlotinib 150 mg/day continuously until disease progression
  Other Names: Tarceva
  Arms: 2

SUMMARY:
The purpose of this study is to assess if the combination of erlotinib and chemotherapy (docetaxel in case of squamous cell NSCLC or pemetrexed in case of other histological types) is superior to erlotinib alone and has acceptable tolerability and safety in the 2nd line treatment of patients with advanced/metastatic non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Open randomized multicenter phase II study in patients in need of 2nd line treatment for advanced/metastatic NSCLC. Efficacy and safety of monotherapy with erlotinib will be compared with combination therapy of erlotinib and chemotherapy. In recent studies it was established that pemetrexed activity is more pronounced in non-squamous NSCLC in comparison to squamous cell carcinoma. Therefore in patients with non-squamous carcinoma pemetrexed will be used. As in second line treatment of NSCLC docetaxel is registered also for usage in patients with squamous cell carcinoma, docetaxel will be used in patients with squamous histology.

Chemotherapy will be limited to 4 courses. Erlotinib will be continued until disease progression or unacceptable toxicity.

Erlotinib as monotherapy will be administered continuously. In combination with chemotherapy, erlotinib will be given from day 2-16 of every course of 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed NSCLC, locally advanced and metastatic disease stage IIIB and IV. Evidence of disease progression after one or two cytotoxic treatment regimens which should have included a platinum agent.
2. Complete recovery from prior chemotherapy side effects to < Grade 2.
3. At least one unidimensional measurable lesion meeting RECIST criteria.
4. ECOG PS 0-2.
5. Age > 18 years.
6. Adequate organ function, including:

   * Adequate bone marrow reserve: ANC > 1.5 x 109/L, platelets > 100 x 109/L.
   * Hepatic: bilirubin <1.5 x ULN, AP, ALT, AST < 1.5 x ULN AP, ALT, and AST <5 x ULN is acceptable if the liver has tumor involvement
   * Renal: calculated creatinin clearance > 40 ml/min based on the Cockcroft-Gault formula.
7. Estimated life expectancy >12 weeks.
8. Male and female patients with reproductive potential must use an approved contraceptive method, if appropriate. Female patients with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.
9. Signed informed consent.
10. Patient compliance and geographical proximity that allow adequate follow up.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with medical risks because of non-malignant disease as well as those with active uncontrolled infection.
3. Documented brain metastases unless the patient has completed local therapy for central nervous system metastases and has been off corticosteroids for at least two weeks before enrollment.
4. Previous treatment with an EGFR-TKI, or in non-squamous histology earlier treatment with pemetrexed and in squamous earlier treatment with docetaxel.
5. Inability to interrupt aspirin or other non-steroidal anti-inflammatory agents for a 5-day period (5 day period for long-acting agents such as piroxicam).
6. Inability or unwillingness to take folic acid, vitamin B-12 supplementation or dexamethasone.
7. Concomitant treatment with any other experimental drug under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2009-03; Primary Completion 2014-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From randomisation to date of first progression or date of death, assessed up to 36 months
  to compare the PFS in the group receiving erlotinib alone versus the patients receiving erlotinib + single agent Progression free survival

SECONDARY OUTCOMES:
Number of Adverse Events | From randomisation to 30 days after EoT all AEs are collected
  to compare relevant toxicity (CTC AE vs 3.0) in the group receiving erlotinib alone versus the patients receiving erlotinib + single agent

CONTACTS AND LOCATIONS:
Overall Officials: Joachim G. Aerts, MD PhD, Study Director — Amphia Ziekenhuis, Breda, The Netherlands; Henk E. Coderington, MD, Study Director — HagaZiekenhuis, The Hague, The Netherlands
Locations (14):
- Netherlands (14):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - VU medisch centrum, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Catharina-Ziekenhuis, Eindhoven
  - Martini Ziekenhuis, Groningen
  - Kennemer Gasthuis, Haarlem
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum Sint Radboud, Nijmegen
  - Maasstad Ziekenhuis, Rotterdam
  - Sint Franciscus Gasthuis, Rotterdam
  - HagaZiekenhuis, The Hague
  - Isala Klinieken, Zwolle

REFERENCES:
- [Result] De Ruysscher D, Dingemans AC, Praag J, Belderbos J, Tissing-Tan C, Herder J, Haitjema T, Ubbels F, Lagerwaard F, El Sharouni SY, Stigt JA, Smit E, van Tinteren H, van der Noort V, Groen HJM. Prophylactic Cranial Irradiation Versus Observation in Radically Treated Stage III Non-Small-Cell Lung Cancer: A Randomized Phase III NVALT-11/DLCRG-02 Study. J Clin Oncol. 2018 Aug 10;36(23):2366-2377. doi: 10.1200/JCO.2017.77.5817. Epub 2018 May 22. PMID 29787357
- [Result] Witlox WJA, Ramaekers BLT, Groen HJM, Dingemans AM, Praag J, Belderbos J, van der Noort V, van Tinteren H, Joore MA, De Ruysscher DKM. Factors determining the effect of prophylactic cranial irradiation (PCI) in patients with stage-III nonsmall cell lung cancer: exploratory subgroup analyses of the NVALT-11/DLCRG-02 phase-III study. Acta Oncol. 2019 Oct;58(10):1528-1531. doi: 10.1080/0284186X.2019.1629016. Epub 2019 Jul 1. No abstract available. PMID 31256737
- [Result] Witlox WJA, Ramaekers BLT, Joore MA, Dingemans AC, Praag J, Belderbos J, Tissing-Tan C, Herder G, Haitjema T, Ubbels JF, Lagerwaard J, El Sharouni SY, Stigt JA, Smit EF, van Tinteren H, van der Noort V, Groen HJM, De Ruysscher DKM. Health-related quality of life after prophylactic cranial irradiation for stage III non-small cell lung cancer patients: Results from the NVALT-11/DLCRG-02 phase III study. Radiother Oncol. 2020 Mar;144:65-71. doi: 10.1016/j.radonc.2019.10.016. Epub 2019 Nov 14. PMID 31733490
- [Derived] Aerts JG, Codrington H, Lankheet NA, Burgers S, Biesma B, Dingemans AM, Vincent AD, Dalesio O, Groen HJ, Smit EF; NVALT Study Group. A randomized phase II study comparing erlotinib versus erlotinib with alternating chemotherapy in relapsed non-small-cell lung cancer patients: the NVALT-10 study. Ann Oncol. 2013 Nov;24(11):2860-5. doi: 10.1093/annonc/mdt341. Epub 2013 Aug 28. PMID 23986090
- See also: Dutch Society of Physicians for Pulmonology and Tuberculosis (NVALT) — http://www.nvalt.nl